CLINICAL TRIAL: NCT04379557
Title: Ablation Index Guided High Power Ablation for Pulmonary Vein Isolation in Patients With Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LESS AF
Record Dates: First submitted 2020-03-17; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2019-11

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High power ablation (Experimental): Ablation Index guided high power ablation (radio frequency energy: Left atrium anterior segment and roof: 40W, Left atrium inferior/posterior: 30W, near esophagus: 25W)
  Interventions: Procedure: Catheter Ablation
- Conventional ablation (Active Comparator): Conventional ablation applying 30-35W strategy for Left atrium anterior segments.
  Interventions: Procedure: Catheter Ablation

INTERVENTIONS:
Procedure: Catheter Ablation — Catheter Ablation is a procedure used to remove or terminate a faulty electrical pathway from sections of the hearts of those who are prone to developing cardiac arrhythmias

SUMMARY:
The investigators will compare the ablation time during pulmonary vein isolation of Ablation Index-guided high power ablation with those with conventional ablation.

Ablation time of conventional group will be used from OPTIMUM study. For secondary outcomes, acute outcomes of pulmonary vein isolation using two different strategies will be compared. During 1 year of follow-up in both groups, atrial fibrillation recurrence will be evaluated. The atrial fibrillation recurrence rate at 1 year after pulmonary vein isolation will be compared between the two groups. In addition, fluoroscopic time, procedure time, and complication rates for the high power ablation group will be compared with those with conventional power.

DETAILED DESCRIPTION:
Ablation Index guided high power ablation will be performed in 70 patients with atrial fibrillation with prospectively and consecutively. A contact force-sensing catheter will be used. Ablation will be performed with point-by-point technique using Visitag automated annotation criteria as below;

Ablation Index(AI) target:

* Anterior/roof : 450 AI
* Anterior near carina area : 500 AI
* Posterior/inferior/carina : 350 AI
* Posterior near carina area : 400 AI
* Area near esophagus :25W, 15sec or 300 AI (no further ablation if esophageal temperature increase more than 39°C)
* Interlesion distance ≤ 4.5mm

VISITAGTM settings

* 2.5mm stability range
* 7 sec stability time
* FOT 25%, 3g force
* Tag size 2mm

Ablation parameters are preset as below;

* RF power range: 40W at anterior/roof, 30W at posterior/inferior, 25W at near esophagus area (decrease power 5W by operator decision)
* Target contact force range: 10-20 g
* Flow rate:
* 8 ml/min for STSF < 30W
* 15 ml/min for STSF ≥ 30W

Acute reconnection will be analysed according to predefined segments.

Subgroup analysis will be performed according to type of AF. Data of patients with paroxysmal atrial fibrillation and persistent atrial fibrillation will be analysed separately, and investigate whether this new ablation strategy is effective in both group of patients. To compare outcomes with OPITMUM phase 2 study, the proportion of patients with paroxysmal and persistent atrial fibrillation would be 75% and 25%. Therefore, 53 patients with paroxysmal atrial fibrillation and 17 patients with persistent atrial fibrillation will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic paroxysmal or persistent AF who failed anti-arrhythmic agents

Exclusion Criteria:

* Patients who had previous ablation for AF
* Patients with left atrial diameter more than 50 mm
* Inability or unwillingness to receive oral anticoagulation with a vitamin K antagonist (VKA) or non-VKA (NOAC) agent
* Known severe left ventricular systolic dysfunction (ejection fraction <35%)
* Pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Ablation time | during procedure
  To compare ablation time of ablation index guided high power ablation for pulmonary vein isolation in patients with atrial fibrillation

SECONDARY OUTCOMES:
residual potential after first pass pulmonary vein encirclement | during procedure
  segment which observed residual potential after first pass pulmonary vein encirclement during procedure (based on predefined pulmonary vein segments)
acute pulmonary vein reconnection | 1 year
  segment which observed early re-connection during procedure (based on predefined pulmonary vein segments) time frame: during procedure (20-30 minutes after pulmonary vein isolation)
any atrial fibrillation/atrial tachycardia recurrence | 1-year after index procedure
  detected by 12-lead electrocardiogram or 24-hour holter monitoring
Total time | during procedure
  Total ablation time, fluoroscopic time, and procedure time
Rate of Complication | 1 year
  Complications associated with procedure.(bleeding, cardiac tamponade, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Euekeun Choi, M.D. Ph.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National university Hostpital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee SR, Park HS, Choi EK, Lee E, Oh S. Acute and long-term efficacy of ablation index-guided higher power shorter duration ablation in patients with atrial fibrillation: A prospective registry. J Arrhythm. 2021 Jul 21;37(5):1250-1259. doi: 10.1002/joa3.12605. eCollection 2021 Oct. PMID 34621423